CLINICAL TRIAL: NCT05923606
Title: State-dependent Modulation of Interactions of Theta and Gamma Rhythms in Working Memory
Brief Title: Modulation of Brain Oscillations Underlying Working Memory
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Hamdi Eryilmaz, PhD, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2023P001479
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Working Memory
Keywords: Working memory; Attention; Theta oscillations; Transcranial Alternating Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Theta-nested gamma tACS applied during passive task epochs (Experimental): Participants will receive single-session administration of tACS during performance of a working memory task. tACS will be applied during fixation periods between consecutive task trials. EEG will be acquired before and immediately after the intervention.
  Interventions: Device: Active tACS
- Theta-nested gamma tACS applied during memory delays (Experimental): Participants will receive single-session administration of tACS during performance of a working memory task. tACS will be applied during memory delays. EEG will be acquired before and immediately after the intervention.
  Interventions: Device: Active tACS
- Gamma tACS applied during memory delays (Experimental): Participants will receive single-session administration of tACS during performance of a working memory task. tACS will be applied during memory delays. The stimulation will be phase locked to the peaks of ongoing theta rhythms of the participant. EEG will be acquired before and immediately after the intervention.
  Interventions: Device: Active tACS
- Placebo tACS applied during task performance (Placebo Comparator): Participants will receive single-session administration of placebo tACS during performance of a working memory task. EEG will be acquired before and immediately after the intervention.
  Interventions: Device: Placebo tACS

INTERVENTIONS:
Device: Active tACS — Active tACS will be administered over the left dorsolateral prefrontal cortex for approximately 25 minutes.
  Arms: Gamma tACS applied during memory delays; Theta-nested gamma tACS applied during memory delays; Theta-nested gamma tACS applied during passive task epochs
Device: Placebo tACS — Placebo tACS will be administered over the left dorsolateral prefrontal cortex for approximately 25 minutes.
  Arms: Placebo tACS applied during task performance

SUMMARY:
This study will use novel transcranial alternating current stimulation (tACS) protocols and electroencephalography (EEG) to modulate and measure brain oscillations that underlie working memory. tACS is a noninvasive method used to modulate the timing and patterns of brain rhythms via weak electric currents passed through electrodes on the scalp.

DETAILED DESCRIPTION:
In this study, healthy adult individuals will perform a spatial working memory task as investigators record scalp EEG before and immediately after undergoing transcranial alternating current stimulation (tACS). Each participant will complete four tACS sessions in randomized order: 1) theta-nested gamma tACS applied during active task periods, 2) theta-nested gamma tACS applied during passive (rest) periods, 3) gamma stimulation applied in phase with ongoing theta oscillations, and 4) placebo tACS. The different stimulation protocols will take place on different days. Therefore, participants will be expected to attend 4 in-person study visits at the Martinos Center for Biomedical Imaging in Charlestown, Massachusetts.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Fluent in English.

Exclusion Criteria:

* History of a neurological/psychiatric disorder
* Current use of psychotropic medications
* Current use of substances and drugs that were shown to affect tES (transcranial electrical stimulation) efficacy (dopamine altering drugs, nicotine, NMDA (N-methyl-D-aspartate) antagonists/agonists, sodium/calcium channel blockers, norepinephrine reuptake inhibitors, GABAergic modulators and selective serotonin reuptake inhibitors)
* Contraindications for tACS (e.g., history of seizures, metallic implants in the head or neck, implanted brain stimulators, vagus nerve stimulators, pacemakers, pregnancy)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Working memory accuracy | 2 hours
  Accuracy of working memory retrieval during a Delayed Match-to-Sample task will be assessed before and during tACS interventions
Working memory accuracy under interference | 2 hours
  Accuracy of working memory retrieval during interference conditions of a Delayed Match-to-Sample task will be assessed before and during tACS interventions.
Theta-gamma cross-frequency coupling | 2 hours
  Cross-frequency coupling between theta band phase and gamma band amplitude will be calculated using the EEG data collected while subjects perform the Delayed Match-to-Sample task before and after tACS interventions.
Fronto-parietal theta phase synchronization | 2 hours
  Phase synchronization in the theta band between frontal and parietal brain regions will be calculated using the EEG data collected while subjects perform the Delayed Match-to-Sample task before and after the tACS interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Hamdi Eryilmaz, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Martinos Center for Biomedical Imaging, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No